CLINICAL TRIAL: NCT01270711
Title: Study on Utilization Of Cabergoline For Compliance With Risk Minimization Activities (SUCRE)
Acronym: SUCRE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A7231030
Record Dates: First submitted 2010-12-09; First posted 2011-01-05 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease; Hyperprolactinemia
Keywords: compliance study; effectiveness study; hyperprolactinemia; Parkinson's disease; retrospective cohort study
MeSH Terms: conditions — Parkinson Disease; Hyperprolactinemia | interventions — Drug Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cabergoline users: cohort of patients, who are treated with cabergoline during the study period ( from January 1st, 2006 to July 1st 2012)
  Interventions: Drug: Study Drug

INTERVENTIONS:
Drug: Study Drug — non interventional study - usage as per usual care

SUMMARY:
The overall goal of this study will be to assess and monitor the adherence to and effectiveness of the new prescribing guidelines for cabergoline.

Specific objectives will be to assess: 1. The indication for use of cabergoline (Parkinson, hyperprolactinemia, other) 2. Prior treatment strategies in patients who start cabergoline treatment for Parkinson's Disease 3. The percentage of cabergoline users who are prescribed doses above 3 mg per day 4. Whether cabergoline users are monitored by echocardiography prior and during treatment. 5. The incidence and prevalence of valvular fibrosis

DETAILED DESCRIPTION:
does not involve random selection

ELIGIBILITY:
Inclusion Criteria:

* Treated with cabergoline during the study period (January 1st, 2006 and will end on July 1st 2012) and identified in one of 6 databases: The Health Information Network, Health Search Database, Integrated Primary Care Information database, PHARMO, Aarhus hospital databases, and the Universitaet Bremen - Bremen Institute for Prevention

Exclusion Criteria:

* Patients with eligibility dates that start after July 1st 2007 (meaning that they would have less than one year of valid data before publication of the results of the EMEA review), will be excluded as well as patients whose eligibility ends before July 1st 2008 (date of SmPC changes).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of patients, who are treated with cabergoline during the study period. This cohort will be divided in new users and prevalent users based on when cabergoline was started. New (incident) users will be all persons who have a first prescription for cabergoline after the date that the change in SPC was made. Prevalent users will be all cohort members who received a cabergoline prescription during the study period but who had also been using cabergoline prior to the change in SPC.
Sampling Method: Non-Probability Sample
Enrollment: 22014 (Actual)
Dates: Start 2010-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7231030&StudyName=Study%20On%20Utilization%20Of%20Cabergoline%20For%20Compliance%20With%20Risk%20Minimization%20Activities%20%28SUCRE%29%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 recruited participants from North, Middle and South Europe and Part 2 from specialized clinical centers in Italy.
Pre-assignment Details: Part 1 assessed adherence (compliance) with prescribing guidelines (PG) by using automated health care data which had information on strength, indication, referrals for echocardiography, recognized reputation in area of drug utilization, safety research. Part 2 assessed effectiveness of PG for cabergoline in participants with Parkinson's disease.
Groups:
- Aarhus [Part 1]: Participants who were registered in Aarhus database and treated with cabergoline during the study period 01 January 2006 through 01 July 2012 (339 weeks) were included. The Aarhus hospital databases comprise clinical and prescription data on the population of Central and the North Denmark Region.
- HSD [Part 1]: Participants who were registered in Health Search Database (HSD) and treated with cabergoline during the study period 01 January 2006 through 01 July 2012 (339 weeks) were included. HSD is a longitudinal observational database that contained data from computer-based participant records of a selected group of general practitioners (GPs) located throughout Italy.
- IPCI [Part 1]: Participants who were registered in Integrated Primary Care Information (IPCI) database and treated with cabergoline during the study period 01 January 2006 through 01 July 2012 (339 weeks) were included. IPCI is a longitudinal observational database that contains data from computer-based participant records of a selected group of GPs throughout the Netherlands.
- PHARMO [Part 1]: Participants who were registered in PHARMO database and treated with cabergoline during the study period 01 January 2006 through 01 July 2012 (339 weeks) were included. PHARMO system linked participants' medical histories to prescription drugs (pharmacy database), diagnostic/therapeutic data from hospitals, clinical lab and pathological findings, GP records and drug histories in hospital throughout the Netherlands.
- THIN [Part 1]: Participants who were registered in The Health Improvement Network (THIN) database and treated with cabergoline during the study period 01 January 2006 through 01 July 2012 (339 weeks) were included. THIN is a database of primary care medical records recorded by the GPs using the vision general practice computer system in the United Kingdom.
- Cabergoline in Pre-SPC Change Period [Part 2]: Participants who started cabergoline treatment for Parkinson's disease prior to the date of the recommended Summary of Product Characteristics (SPC) change, 26 June 2008 (Week 130) and stopped treatment before the recommended change to the SPC.
- Cabergoline in Post- SPC Change Period [Part 2]: Participants who started cabergoline treatment for Parkinson's disease after the date of the recommended SPC change, 26 June 2008 (Week 130).
- Cabergoline in Cross-SPC Change Period [Part 2]: Participants who started cabergoline treatment for Parkinson's disease prior to date of the recommended SPC change, 26 June 2008 (Week 130) and continued treatment after the recommended change to the SPC.
Period: Part 1: Compliance
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1] | Cabergoline in Pre-SPC Change Period [Part 2] | Cabergoline in Post- SPC Change Period [Part 2] | Cabergoline in Cross-SPC Change Period [Part 2]
Started | 7537 | 6580 | 326 | 5486 | 2024 | 0 | 0 | 0
Completed | 7537 | 6580 | 326 | 5486 | 2024 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Effectiveness
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1] | Cabergoline in Pre-SPC Change Period [Part 2] | Cabergoline in Post- SPC Change Period [Part 2] | Cabergoline in Cross-SPC Change Period [Part 2]
Started | 0 | 0 | 0 | 0 | 0 | 11 | 2 | 48
Completed | 0 | 0 | 0 | 0 | 0 | 11 | 2 | 48
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study population included all participants who were treated with cabergoline, registered in one of the databases and those recruited from specialized clinical centers in Italy for Parkinson’s disease during the study period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1] | Cabergoline in Pre-SPC Change Period [Part 2] | Cabergoline in Post- SPC Change Period [Part 2] | Cabergoline in Cross-SPC Change Period [Part 2] | Total
Number analyzed (Participants) | 7537 | 6580 | 326 | 5486 | 2024 | 11 | 2 | 48 | 22014
Age, Customized [Mean (Standard Deviation); unit: years] — Age is stratified by Part 1 and Part 2, in Part 1 age is further stratified by indication, cabergoline use for prolactin reduction indication (ATC [Anatomical Therapeutic Code] G02CB03) and neurological indication (ATC N04BC06).
  years
    Part 1, Compliance: G02CB03 | 33.6 (10.7) | 39.0 (12.3) | 42.1 (14.0) | 41.3 (15.8) | 47.1 (16.2) | NA (NA) — This arm is used for Part 2, Effectiveness. | NA (NA) — This arm is used for Part 2, Effectiveness. | NA (NA) — This arm is used for Part 2, Effectiveness. | 40.8 (14.8)
    Part 1, Compliance: N04BC06 | 66.4 (13.2) | 73.1 (11.3) | NA (NA) — Data not reported as no participants were included in this arm for specified indication. | NA (NA) — Data not reported as no participants were included in this arm for specified indication. | 69.7 (13.6) | NA (NA) — This arm is used for Part 2, Effectiveness. | NA (NA) — This arm is used for Part 2, Effectiveness. | NA (NA) — This arm is used for Part 2, Effectiveness. | 70.4 (13.0)
    Part 2, Effectiveness | NA (NA) — This arm is used for Part 1, Compliance. | NA (NA) — This arm is used for Part 1, Compliance. | NA (NA) — This arm is used for Part 1, Compliance. | NA (NA) — This arm is used for Part 1, Compliance. | NA (NA) — This arm is used for Part 1, Compliance. | 62.7 (5.6) | 58.7 (8.5) | 63.7 (13.9) | 63.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7429 | 6180 | 288 | 5180 | 1468 | 2 | 0 | 13 | 20560
  Male | 108 | 400 | 38 | 306 | 556 | 9 | 2 | 35 | 1454

OUTCOME MEASURES:

1. Primary Outcome: Number of Cabergoline Prescriptions by Database and Indication: Year 1
Description: Cabergoline prescriptions were stratified by indications per year. Indications were coded using Anatomical Therapeutic Code (ATC) which included G02CB03 for prolactin reduction indication and N04BC06 for neurological indication.
Time Frame: Year 1 (Year 2006)
Population: Study population included all participants who were registered in one of the databases and were treated with cabergoline during the study period. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 81 | 854 | 5 | 277 | 370
prescriptions
  G02CB03 | 17 | 1782 | 6 | 293 | 198
  N04BC06 | 87 | 1483 | 0 | 0 | 577

2. Primary Outcome: Number of Cabergoline Prescriptions by Database and Indication: Year 2
Description: as for outcome 1
Time Frame: Year 2 (Year 2007)
Population: as for outcome 1
Measure: Number; unit: prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1446 | 1475 | 31 | 1231 | 756
prescriptions
  G02CB03 | 1925 | 3616 | 64 | 2698 | 3537
  N04BC06 | 741 | 2139 | 0 | 0 | 3325

3. Primary Outcome: Number of Cabergoline Prescriptions by Database and Indication: Year 3
Description: as for outcome 1
Time Frame: Year 3 (Year 2008)
Population: as for outcome 1
Measure: Number; unit: prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1469 | 1089 | 59 | 1081 | 279
prescriptions
  G02CB03 | 2098 | 3493 | 152 | 2621 | 3556
  N04BC06 | 507 | 807 | 0 | 0 | 1656

4. Primary Outcome: Number of Cabergoline Prescriptions by Database and Indication: Year 4
Description: as for outcome 1
Time Frame: Year 4 (Year 2009)
Population: as for outcome 1
Measure: Number; unit: prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1539 | 1146 | 87 | 1039 | 220
prescriptions
  G02CB03 | 2260 | 3629 | 226 | 2684 | 3240
  N04BC06 | 306 | 463 | 0 | 0 | 1119

5. Primary Outcome: Number of Cabergoline Prescriptions by Database and Indication: Year 5
Description: as for outcome 1
Time Frame: Year 5 (Year 2010)
Population: as for outcome 1
Measure: Number; unit: prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1539 | 1050 | 88 | 1005 | 201
prescriptions
  G02CB03 | 2395 | 3793 | 283 | 2752 | 3170
  N04BC06 | 201 | 274 | 0 | 0 | 981

6. Primary Outcome: Number of Cabergoline Prescriptions by Database and Indication: Year 6
Description: as for outcome 1
Time Frame: Year 6 (Year 2011)
Population: as for outcome 1
Measure: Number; unit: prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1463 | 966 | 56 | 853 | 198
prescriptions
  G02CB03 | 2286 | 3686 | 183 | 2660 | 3212
  N04BC06 | 141 | 143 | 0 | 0 | 859

7. Primary Outcome: Percentage of Second-line Prescriptions of Cabergoline for Parkinson's Disease Indications: Year 1
Description: Changes to the Summary of Product Characteristics (SPC) included that the cabergoline should be used for Parkinson's disease only in participants who had already taken or cannot take other treatments, which was as second line therapy. Second-line use restriction did not apply to the hyperprolactinemia indication, for which cabergoline was considered a first-time therapy. Percentage of second-line prescriptions of a total number of prescriptions for cabergoline during a respective year for the neurological indication was reported.
Time Frame: Year 1 (Year 2006)
Population: Study population: participants registered in one of databases and were treated with cabergoline during study period. Data not reported for IPCI and PHARMO databases because no information was retrieved for second-line prescriptions of cabergoline for Parkinson's disease. 'N' (number of participants analyzed)=participants evaluable for this measure.
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 64 | 231 | 242
percentage of prescriptions | 0 | 0 | 0

8. Primary Outcome: Percentage of Second-line Prescriptions of Cabergoline for Parkinson's Disease Indications: Year 2
Description: as for outcome 7
Time Frame: Year 2 (Year 2007)
Population: as for outcome 7
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 49 | 139 | 75
percentage of prescriptions | 4 | 10 | 10

9. Primary Outcome: Percentage of Second-line Prescriptions of Cabergoline for Parkinson's Disease Indications: Year 3
Description: as for outcome 7
Time Frame: Year 3 (Year 2008)
Population: as for outcome 7
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 13 | 18 | 28
percentage of prescriptions | 20 | 39 | 23

10. Primary Outcome: Percentage of Second-line Prescriptions of Cabergoline for Parkinson's Disease Indications: Year 4
Description: as for outcome 7
Time Frame: Year 4 (Year 2009)
Population: as for outcome 7
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 9 | 4 | 20
percentage of prescriptions | 7 | 22 | 12

11. Primary Outcome: Percentage of Second-line Prescriptions of Cabergoline for Parkinson's Disease Indications: Year 5
Description: as for outcome 7
Time Frame: Year 5 (Year 2010)
Population: as for outcome 7
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 6 | 4 | 13
percentage of prescriptions | 18 | 43 | 21

12. Primary Outcome: Percentage of Second-line Prescriptions of Cabergoline for Parkinson's Disease Indications: Year 6
Description: Changes to the Summary of Product Characteristics (SPC) in April 2007 included that the cabergoline should be used for Parkinson's disease only in participants who have already taken or cannot take other treatments, that is as second line therapy. Second-line use restriction did not apply to the hyperprolactinemia indication, for which cabergoline is considered a first-time therapy. Percentage of second-line prescriptions of a total number of prescriptions for cabergoline during a respective year for the neurological indication was reported.
Time Frame: Year 6 (Year 2011)
Population: as for outcome 7
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 2 | 2 | 6
percentage of prescriptions | 11 | 67 | 0

13. Primary Outcome: Percentage of Cabergoline Prescriptions for Dosages Greater Than 3 Milligram (mg) Per Day: Year 1
Description: The Committee for Medicinal Products for Human Use (CHMP) recommended that the prescribing information for cabergoline should be updated to include: a reduction of the maximum recommended dose to 3 mg per day. To evaluate compliance with the new prescription guidelines, it was assessed whether the dose exceeded 3 mg per day during the study period.
Time Frame: Year 1 (Year 2006)
Population: as for outcome 1
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 81 | 854 | 5 | 277 | 370
percentage of prescriptions | 0 | 5 | 0 | 0 | 17

14. Primary Outcome: Percentage of Cabergoline Prescriptions for Dosages Greater Than 3 Milligram (mg) Per Day: Year 2
Description: as for outcome 13
Time Frame: Year 2 (Year 2007)
Population: as for outcome 1
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1446 | 1475 | 31 | 1231 | 756
percentage of prescriptions | 0.2 | 5 | 2 | 0 | 13

15. Primary Outcome: Percentage of Cabergoline Prescriptions for Dosages Greater Than 3 Milligram (mg) Per Day: Year 3
Description: as for outcome 13
Time Frame: Year 3 (Year 2008)
Population: as for outcome 1
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1469 | 1089 | 59 | 1081 | 279
percentage of prescriptions | 0 | 3 | 5 | 0 | 7

16. Primary Outcome: Percentage of Cabergoline Prescriptions for Dosages Greater Than 3 Milligram (mg) Per Day: Year 4
Description: as for outcome 13
Time Frame: Year 4 (Year 2009)
Population: as for outcome 1
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1539 | 1146 | 87 | 1039 | 220
percentage of prescriptions | 0 | 2 | 1 | 0 | 5

17. Primary Outcome: Percentage of Cabergoline Prescriptions for Dosages Greater Than 3 Milligram (mg) Per Day: Year 5
Description: as for outcome 13
Time Frame: Year 5 (Year 2010)
Population: as for outcome 1
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1539 | 1050 | 88 | 1005 | 201
percentage of prescriptions | 0 | 3 | 1 | 0 | 2

18. Primary Outcome: Percentage of Cabergoline Prescriptions for Dosages Greater Than 3 Milligram (mg) Per Day: Year 6
Description: as for outcome 13
Time Frame: Year 6 (Year 2011)
Population: as for outcome 1
Measure: Number; unit: percentage of prescriptions
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1]
Number analyzed (Participants) | 1463 | 966 | 56 | 853 | 198
percentage of prescriptions | 0 | 1 | 0 | 0 | 2

19. Primary Outcome: Total Number of Echocardiography Examinations in Cabergoline Users
Description: The CHMP recommended that the prescribing information for cabergoline should be updated to include: a warning stating that participant must be monitored for signs of cardiac valve fibrosis with echocardiography before treatment is started and regularly (every 6 months) during treatment. To evaluate effectiveness with the new prescription guidelines, it was assessed whether cabergoline users were monitored by echocardiography.
Time Frame: Baseline (Week 1) up to Week 339
Population: Study population included all participants who were recruited from specialized clinical centers in Italy and treated with cabergoline for Parkinson's disease during the study period.
Measure: Number; unit: echocardiography examinations
Groups:
- Cabergoline in Cross-SPC Change Period [Part 2]: Participants who started cabergoline treatment for Parkinson's disease prior to SPC change (26 June 2008) and continued treatment after the recommended change to the SPC.
Arm/Group | Cabergoline in Pre-SPC Change Period [Part 2] | Cabergoline in Post- SPC Change Period [Part 2] | Cabergoline in Cross-SPC Change Period [Part 2]
Number analyzed (Participants) | 11 | 2 | 48
echocardiography examinations | 11 | 3 | 68

20. Primary Outcome: Incidence of Valvular Fibrosis
Description: Incidence of valvular fibrosis was calculated as number of participants with documented valvulopathy during cabergoline treatment and absence of any valve damage at baseline divided by number of participants without any valve damage at baseline and at least 1 additional echocardiography examination during follow-up while on cabergoline treatment. Percentage of participants with valvular fibrosis are reported.
Time Frame: Baseline (Week 1) up to Week 339
Population: Study population:all participants recruited from specialized clinical centers in Italy and treated with cabergoline for Parkinson's disease during study period.
Measure: Number; unit: percentage of participants
Arm/Group | Cabergoline in Pre-SPC Change Period [Part 2] | Cabergoline in Post- SPC Change Period [Part 2] | Cabergoline in Cross-SPC Change Period [Part 2]
Number analyzed (Participants) | 11 | 2 | 48
percentage of participants | 100 | 0 | 57.1

21. Primary Outcome: Prevalence of Valvular Fibrosis
Description: Prevalence of valvular fibrosis was calculated as number of participants with documented valvulopathy during cabergoline treatment divided by number of participants with at least 1 echocardiography examination. Percentage of participants with valvular fibrosis are reported.
Time Frame: Baseline (Week 1) up to Week 339
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Cabergoline in Pre-SPC Change Period [Part 2] | Cabergoline in Post- SPC Change Period [Part 2] | Cabergoline in Cross-SPC Change Period [Part 2]
Number analyzed (Participants) | 11 | 2 | 48
percentage of participants | 57.2 | 50.0 | 55.9

ADVERSE EVENTS:
Description: This retrospective study used participant-level electronic health related databases, in which adverse events (AEs) were not reportable as an individual AE report because an AE data for individual participant was not available.
Arm/Group | Aarhus [Part 1] | HSD [Part 1] | IPCI [Part 1] | PHARMO [Part 1] | THIN [Part 1] | Cabergoline in Pre-SPC Change Period [Part 2] | Cabergoline in Post- SPC Change Period [Part 2] | Cabergoline in Cross-SPC Change Period [Part 2]
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Results not reported for Year 2012 (Year 7) since several databases did not contribute data for Year 7 and amount of person-time of follow-up dropped in all databases. Designation of primary and secondary endpoints was based on study team's input.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.